CLINICAL TRIAL: NCT01352403
Title: Severe Obesity: Bariatric Surgery vs. Life-Style-Intervention Wurzburg Adipositas Study - WAS
Brief Title: Severe Obesity: Bariatric Surgery vs. Life-Style-Intervention
Acronym: WAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wuerzburg (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Martin Fassnacht, Chair of Department of Endocrinology and Diabetology, University of Wuerzburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-005054-20
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Obesity; Cardiac Function; Quality of Life
Keywords: obesity; bariatric surgery; gastric bypass; life style intervention; cardiac function
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychotherapy-enhanced lifestyle intervention (PELI) (Other): Intensive lifestyle intervention over 12 months including medically supervised dietary counseling and physical activity enhanced by a psychotherapeutic intervention
  Interventions: Behavioral: Psychotherapy-enhanced lifestyle intervention
- Roux-en-Y-gastric bypass (RYGB) (Other): Laparoscopic Roux-en-Y gastric bypass surgery
  Interventions: Procedure: Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass
  Arms: Roux-en-Y-gastric bypass (RYGB)
Behavioral: Psychotherapy-enhanced lifestyle intervention
  Arms: Psychotherapy-enhanced lifestyle intervention (PELI)

SUMMARY:
The purpose of this study is to investigate the effects of weight loss induced by gastric bypass surgery in comparison to a psychotherapy-enhanced lifestyle intervention on cardiopulmonary performance and quality of life in patients with morbid obesity.

DETAILED DESCRIPTION:
Obesity is a rapidly emerging health problem and an established risk factor for cardiovascular diseases. Bariatric surgery profoundly reduces body weight and mitigates sequelae of obesity. Especially randomized trials comparing the effects of bariatric surgery to conservative treatment in concerns of cardiac function are still lacking.

The randomized WAS trial compares the effects of Roux-en-Y gastric bypass (RYGB) versus psychotherapy-supported lifestyle modification in morbidly obese patients. The co-primary endpoint addresses 1-year changes in cardiovascular function (peak VO2 during cardiopulmonary exercise testing) and quality of life (Short-Form-36 physical functioning scale). Prior to randomization, all included patients underwent a multimodal anti-obesity treatment for 6-12 months. Thereafter, patients were randomized and followed through month 12 to collect primary endpoints. Afterwards, patients in the lifestyle group could opt for surgery, and final visit was scheduled for all patients 24 months after randomization.

The study was initially designed in 2008 as part of several interdisciplinary studies for a targeted grant and received a positive vote from the responsible ethics committee.

Prior the actual start of the study in July 2011, the initial study protocol and the patient informed consent were updated and further specified. This amendment was submitted to the Ethics Committee on June 9, 2011, with a positive vote on June 30, 2011 (Amendment 1).

An Amendment 2 was submitted to Ethics Committee on 08.10.2014 (positive vote 16.12.2014) to adjust randomization (previously 1:1 to the two study arms) for an unequal drop-out rate in the two study arms with higher rate in the intensified lifestyle modification. In addition, few secondary endpoints were adapted and the role of the principal investigator changed from Prof. Stefan Frantz to Prof. Martin Fassnacht.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* BMI >40 kg/m2 or BMI >35 kg/m2 with severe comorbidities
* Indication for Roux-en-Y gastric bypass surgery
* Ability to perform cardiopulmonary exercise testing (CPET)
* Written informed consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Unstable angina pectoris
* Life expectancy <12 months
* Endocrine or psychiatric disorder as cause of obesity
* Systemic glucocorticoid treatment (with exception of glucocorticoid replacement therapy)
* Abuse of drugs or alcohol within the last 5 years
* Inability to attend regular study visits for logistic reasons
* Participation in competing trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-07-04 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Change of peak VO2 to assess cardiorespiratory performance | 12 months after surgery / lifestyle intervention
  Change of peak V O2 (measured in ml/min/kg bw) in cardiopulmonary exercise testing (CPET)
Change in physical functioning scale (PFS) of the SF-36 to assess quality of life | 12 months after surgery / lifestyle intervention
  Change of quality of life measured with physical functioning scale (PFS) of the SF-36 questionnaire (Short Form health survery 36). The score ranges from 0-100 and higher values correspond to better quality of life.

SECONDARY OUTCOMES:
Change in health related quality of life (other domains than physical functioning scale) | 12 and 24 months after bariatric surgery / lifestyle intervention
  Change in quality of life (using Short Form (SF-36) health survey 36). The score ranges from 0-100 and higher values correspond to better quality of life.
Change in left ventricular mass (index) | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment with echocardiography (g and g/m^2 body surface area)
Changes in left atrial dimensions | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment with echocardiography (left atrial enddiastolic volume (mm^3), left atrial enddiastolic diameter (mm))
Changes in left ventricular dimensions | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment with echocardiography (left ventricular enddiastolic volume (mm^3), left ventricular enddiastolic diameter (mm))
Change in left ventricular systolic function | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment with echocardiography (left ventricular ejection fraction (%), longitudinal strain)
Change in prevalence of left ventricular diastolic dysfunction | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment with echocardiography (Defined as reduced LVEF, LV hypertrophy, or LV dilation, as well as if three out of the following four criteria were fulfilled 77: LA dilation, average E/e' >14, lateral e' <0.1 m/s or septal e' <0.07 m/s, tricuspid regurgitation maximal flow velocity >2.8 m/s)
Change in physical performance | 12 and 24 months after bariatric surgery / lifestyle intervention
  Distance (m) achieved in the 6 minute walk test
Change in brain morphology | 12 and 24 months after bariatric surgery / lifestyle intervention
  Structural MRI of the brain to assess change in grey matter volume of the cerebellum (compared to normal weight controls)
Change in brain activity | 12 and 24 months after bariatric surgery / lifestyle intervention
  Functional MRI of the brain to assess activation to high caloric food stimuli in obese patients in insula and anterior cingulate gyrus (compared to normal weight controls)
Change in brain oxygenation | 12 and 24 months after bariatric surgery / lifestyle intervention
  Functional near-infrared spectroscopy (fNIRS) with assessment of frontal cortical oxygenation during Verbal Fluency Test and Trail Making Test and assessment of low frequency oscillations in resting state (in comparison to normal weight controls)
Change in left ventricular function | 12 and 24 months after bariatric surgery / lifestyle intervention
  Cardiac MR imaging with analysis of left ventricular function (left ventricular ejection fraction, %)
Change in cardiac lipid content | 12 and 24 months after bariatric surgery / lifestyle intervention
  Cardiac MR imaging with spectroscopy to measure cardiac lipid content (% fat content)
Change in depressed mood | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment of depressed mood using Patient Health Questionnaire 9 (PHQ-9). The score ranges from 0-27, higher values correspond to more pronounced depressive symptoms.
Change in depression | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment of depressed mood using Beck's Depression Inventory (BDI-II). The score ranges from 0-63, higher values correspond to more pronounced depressive symptoms.
Change in liver stiffness | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment of liver stiffness using transient elastography (kPa)
Change in liver triglyceride content | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment of liver triglyceride content with MR spectroscopy (% liver fat)
Change in burden of comorbidities (type 2 diabetes mellitus) | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment of type 2 diabetes by predefined criteria. If the patient fulfils one of the following criteria, he/she would count as diabetic patient: fasting blood sugar level >= 126mg/dl, A1c => 6.5%, glucose of >=200 mg/dl 2hours in oral glucose tolerance test, or use of at least one antidiabetic medication.
Change in burden of comorbidities (arterial hypertension) | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment of arterial hypertension according to predefined criteria. If the patient fulfils one of the following criteria, he/she would count as antihypertensive: systolic blood pressure >= 140mmHg, diastolic blood pressure >= 90mmHg, or use of at least one antihypertensive drug.
Change in burden of comorbidities (dyslipidemia) | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment of dyslipidemia according to predefined criteria (depending on values for fasting triglycerides and ldl-cholesterol, lipid lowering medication)
Change in NYHA functional class | 12 and 24 months after bariatric surgery / lifestyle intervention
  Assessment of NYHA functional class (NYHA I-IV, a higher class meaning more dyspnea)

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital, University of Wuerzburg, Würzburg, Bavaria, Germany

REFERENCES:
- [Background] Koschker AC, Warrings B, Morbach C, Seyfried F, Rickert N, Jung P, Geier A, Dischinger U, Krauthausen M, Herrmann MJ, Stier C, Frantz S, Malzahn U, Stork S, Fassnacht M. Cardio-psycho-metabolic outcomes of bariatric surgery: design and baseline of the WAS trial. Endocr Connect. 2022 Feb 9;11(2):e210338. doi: 10.1530/EC-21-0338. PMID 35015697